CLINICAL TRIAL: NCT03601273
Title: Bariatric Embolization Trial for the Obese Nonsurgical
Acronym: BET-ON
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Calgary Adult Bariatric Surgery Clinic (Other); Peter Lougheed Center, Mayfair Diagnostics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB17-0610
Record Dates: First submitted 2018-07-09; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Obesity; Weight Loss; Body Weight; Morbid Obesity
Keywords: left gastric artery embolization; bariatric embolization; interventional radiology; obesity; morbid obesity; weight loss
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Left gastric artery embolization — 450-micron Embozene microparticles will be used intraarterially to occlude the left gastric artery and its branches.
  30-day post-embolization endoscopic biopsy
  Other Names: bariatric embolization

SUMMARY:
The purpose of this study is to assess the safety profile of bariatric embolizations and confirm published reports of sustained post-procedural weight loss, and pathologically assess post-procedural metabolic effects.

DETAILED DESCRIPTION:
Since 2003, the proportion of Canadians who were obese has increased 17.5%. Obesity is ranked as the fifth leading risk for mortality globally. Obesity has been strongly linked to numerous comorbidities, including type II diabetes, hyperlipidemia, hypertension, obstructive sleep apnea, heart disease, stroke, asthma, cancer, and depression.

The pathophysiology of obesity is complex and inadequately understood. Nevertheless, an energy imbalance is fundamentally at fault. As recently as 1996, ghrelin, the hormonal stimulus for hunger was identified. Further research has revealed that ghrelin, predominantly produced in the fundus of the stomach, stimulates appetite and increases serum concentrations of growth hormone, adrenocorticotropic hormone, cortisol, prolactin, and glucose.

Congruously, the complexity of obesity is reflected in the efficacy of modern therapy. Treatment for obesity lies along a spectrum of available modalities beginning with diet modification, exercise therapy, pharmacotherapy, and surgery. Despite initial positive results, diet and exercise frequently prove futile for long-term management of weight loss. Likewise, it is uncommon for diabetic remission to be achieved through pharmaco-therapeutic agents, most of the medications designed to stabilize and improve diabetic control. This has led to the advent of interventional treatment for these conditions.

Bariatric surgery is the current gold-standard in the treatment of morbid obesity with recent evidence revealing that bariatric surgery is more effective than medical treatment for the long-term control of obese patients with type 2 diabetes. It is postulated that in addition to the restrictive effects associated with bariatric surgery, resection or disruption of the ghrelin producing regions of the stomach may play a significant role in eventual weight loss.

The primary source of blood flow to the fundus of the stomach, where the majority of ghrelin-producing cells are found, is the left gastric artery. This artery is commonly accessed percutaneously for the management of refractory upper gastrointestinal bleeding. Embolizations are typically well tolerated, therefore, it has been purported that selective embolization of this artery could induce adequate ischemia to the fundus resulting in a rapid decrease in ghrelin-producing cells along with its neurological and metabolic effects.

In 2007, Arepally et al reported a minimally-invasive method of destroying ghrelin-producing cells in a porcine model. With mixed success, Arepally was able to demonstrate a correlation between left gastric artery embolizations, weight loss, and fluctuations in ghrelin levels. Propagation of his efforts was performed by Bawudun et al, utilizing a liquid sclerosant and 500-700-mm polyvinyl alcohol (PVA) particles as embolic agents, Bawudun was able to demonstrate significant decreases in ghrelin and body weight measurements in the experimental arms in a canine model. Subsequently, Paxton, et al. demonstrated lowered ghrelin levels and reduced weight gain utilizing 40-micron microsphere particle embolizations in a similar porcine model no duodenal upregulation for ghrelin was found. These studies also revealed potential complications including non-target embolization, frank gastric ulcerations, and gastritis.

Following these preclinical animal studies, Gunn and Oklu performed a small retrospective study of patients who underwent a left gastric artery embolization for upper gastrointestinal bleeds. The results, although limited, revealed significant weight loss amongst the experimental group as compared with the control (patients who underwent embolization for upper gastrointestinal bleeds without left gastric artery selection). Kipshidze et al reported significant weight loss amongst all five patients who underwent the first-in-human prospective left gastric artery embolization trial utilizing 300-500 µm microspheres. Human trials have resulted in few reported complications, namely minor pyrosis and indigestion. The safety profile of the procedure is well reported given that elective left gastric artery embolizations are offered to stable patients with refractory non-variceal bleeds. Case reports have reported on the uncommon instances of hepatic infarction, gastric infarction, gastric volvulus, and arterial rupture.

The momentum behind this procedure has led to the design and implementation of two phase I clinical trials [Gastric Artery Embolization Trial for the Lessening of Appetite Nonsurgically (GET LEAN) and Bariatric Embolization of Arteries for the Treatment of Obesity (BEAT Obesity)] which sought to demonstrate the safety profile of left gastric artery embolizations and demonstrate post-procedural weight loss.

Results have been promising with weight loss and safety demonstrated in both trials.

Minor complications included post-procedural nausea, vomiting, and mild epigastric discomfort which was treated with oral proton pump inhibitors (PPIs) following administration of one course of intravenous (IV) PPIs. 3 asymptomatic gastric ulcers were identified on post-procedural endoscopy however these resolved within 1 month (a 1-month endoscopy was performed).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are bariatric surgical candidates; however, have refused surgery.
* BMI >40
* BMI between 35 and 40 with medical comorbidities
* Patients who meet criteria for medical management of obesity with BMI ≥ 35
* Age ≥ 18 years
* Willing, able and mentally competent to provide written informed consent

Exclusion Criteria:

* Age less than 18 years of age
* Inability to lay supine on an angiographic table <500lbs due to table weight limits
* Inappropriate anesthesia risk as determined by certified anesthesia provider.
* Presence of a contraindication to endovascular therapy
* Major surgery within the past eight weeks
* Previous gastric, pancreatic, hepatic and splenic surgery
* Previous radiation therapy to the left or right upper quadrant
* Previous gastric, hepatic, or splenic embolization
* Any history of portal venous hypertension
* Severe renal impairment resulting in unacceptable risk of contrast-induced nephropathy
* Pregnant or intend to become pregnant within one year
* History of severe bleeding disorder (platelet count less than 40,000)
* Allergy to materials in the embolic agents
* Enrolled in another study
* Any patient who has a history of allergic reaction to iodinated contrast
* Abnormal baseline gastric emptying study
* Patients taking anti-coagulants (anti-platelets fine)
* Patients currently taking or requiring chronic use of non steroidal anti-inflammatory drugs (NSAID) or steroid medications
* Patients with any chronic upper gastrointestinal complaints such as pain, nausea or vomiting
* Patients with any history of peptic ulcer disease
* Patients with any indication of gastrointestinal bleeding as documented by positive stool guaiac and complete blood count with abnormalities.
* Subjects with mesenteric atherosclerotic disease or abdominal angina should be excluded due to safety concerns.
* Patients with known aortic disease, such as dissection or aneurysm
* Patients with comorbidities such as cancer
* Patients with any abnormality on their baseline esophagogastroduodenoscopy (EGD)
* Patients with a CT Angiogram demonstrating an anatomical variant in left gastric artery anatomy
* Patients with any contraindications for monitored anesthesia care or general surgery
* Patients with secondary causes of obesity such as Cushing's disease, hypothyroidism, or abnormal testosterone readings
* Patients with active substance abuse or alcoholism
* Patients with defined noncompliance with previous medical care
* Patients with certain psychiatric disorders such as schizophrenia, borderline personality disorder, and uncontrolled depression, and mental/cognitive impairment that limits the individual's ability to understand the proposed therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 5 years
  Safety outcomes involving the use of left gastric artery embolization

SECONDARY OUTCOMES:
Change in Body mas index (BMI) | 5 years
  kg/m2
Percentage estimated body weight loss (EBWL) | 5 years
Change in concentration of Ghrelin-producing cells | 30 days post-operative
  Concentration of Ghrelin-producing cells pre-embolization obtained through endoscopic biopsy and measured by cells per milliliter, will be subtracted from the concentration of Ghrelin-producing cells obtained post-embolization from endoscopic biopsy. This value will be converted into a percentage change and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Darshan Bakshi, MD, Principal Investigator — University of Calgary; Oliver Halliwell, MD, Study Director — University of Calgary; Emeka Nzekwu, MD, Study Director — University of Calgary

IPD SHARING:
Plan to Share IPD: Undecided